CLINICAL TRIAL: NCT02121938
Title: Dynamics of the Microbiome in the Premature Infant
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00051659
Record Dates: First submitted 2014-04-21; First posted 2014-04-24 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2016-06

CONDITIONS: Infection
Keywords: Very Low Birth Weight (VLBW); Microbiome
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, stool, serum, breastmilk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- very low birth weight infants: Very low birth weight infants weighing 1500 grams at birth or less

SUMMARY:
The purpose of the study is to describe the dynamics of the microbiome in the premature infant as a means to adapt the premature infant gut to affect better health outcomes.

DETAILED DESCRIPTION:
The study team will collect samples of blood and stool from preterm infants once a week from the first week of life until 8 weeks after delivery. Blood samples will be collected from left over blood that is being collected for clinical management. No extra blood draws will be done for research purposes only. Samples of leftover breast milk will be collected once weekly from the first week of life until 8 weeks after delivery.

While the baby is in the hospital the study team will collect information about the growth and development as well as events that happen during their intensive care nursery (ICN) hospitalization.

In addition, blood and stool will be collected, as well as information about the growth when the infant returns to the Duke Special Infant Care Clinic for developmental check-ups at 6 and 12 months of age. The blood will be approximately 1 teaspoon (5 milliliters) and will be done at the same time that labs for clinical management are being done.

A single maternal blood sample (approximately 2 teaspoons) and stool sample will be collected after delivery. Information will also be collected from the medical record.

ELIGIBILITY:
Inclusion Criteria:

* 1500 grams or less at birth
* infants without genetic diseases or gross anomalies
* mother has to be planning on providing breast milk to the infant

Exclusion Criteria:

* infants with genetic diseases or gross anomalies
* parents who are not willing to give consent

Ages: 1 Hour to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very low birth weight infants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
antigen identification of the infant microbiome over the first year of life | Week 1
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.
antigen identification of the infant microbiome over the first year of life | Week 2
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.
antigen identification of the infant microbiome over the first year of life | Week 3
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.
antigen identification of the infant microbiome over the first year of life | Week 4
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.
antigen identification of the infant microbiome over the first year of life | Week 5
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.
antigen identification of the infant microbiome over the first year of life | Week 6
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.
antigen identification of the infant microbiome over the first year of life | Week 7
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.
antigen identification of the infant microbiome over the first year of life | Week 8
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.
antigen identification of the infant microbiome over the first year of life | 6 months
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.
antigen identification of the infant microbiome over the first year of life | 12 months
  The investigators immediate goal is to identify antigens of the preterm infant microbiome that are recognized by natural and adaptive antibodies and determine how mucosal and serologic antibody responses alter the dynamics of secondary intestinal colonization.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Seed, MD PhD, Principal Investigator — Duke Univeristy
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States